CLINICAL TRIAL: NCT01007864
Title: Influence of the Non-Ergot Dopamine Agonist Piribedil on Vigilance and Cognitive Function in Patients With Parkinson's Disease Compared to Other Oral Non-Ergot Dopamine Agonists
Brief Title: Influence of Piribedil (Clarium®) on Vigilance and Cognitive Function in Patients With Parkinson's Disease Compared to Other Non-Ergot Dopamine Agonists
Acronym: PIVICOG-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Desitin Arzneimittel GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIR-007/K
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-04

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson; piribedil; vigilance; dopamine agonist; cognition
MeSH Terms: conditions — Parkinson Disease | interventions — Piribedil; Loratadine; Pramipexole; ropinirole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- piribedil (Experimental)
  Interventions: Drug: piribedil
- pramipexole or ropinirole (Active Comparator)
  Interventions: Drug: pramipexole or ropinirole

INTERVENTIONS:
Drug: piribedil — Oral application of piribedil at an equivalent dose of pramipexole or ropinirole according to a defined equivalence scheme (dose range 100 - 300 mg per day) for 11 weeks.
  Other Names: Clarium®
  Arms: piribedil
Drug: pramipexole or ropinirole — continuation of pre-study treatment regimen
  Arms: pramipexole or ropinirole

SUMMARY:
The purpose of this clinical trial is to investigate the effects of the non-ergot dopamine agonist piribedil on vigilance and cognitive performances in patients with Parkinson's disease in comparison with other oral non-ergot dopamine agonists.

It should be tested whether piribedil is superior to continued pramipexole or ropinirole treatment regarding improvement of reduced vigilance and cognitive performance in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Treatment of motor symptoms associated with PD by non-ergot dopamine agonists has been proven to be effective, both as monotherapy and in combination with levodopa. Non-motor symptoms like cognitive or sleep-related disorders and disturbed vigilance, however, are common in PD and can significantly worsen health and quality of life of the patient and family members. Some of these non-motor symptoms may also be caused by the antiparkinsonian medication per se. The Committee for Proprietary Medicinal Products (CPMP) initiated a review of dopamine agonists in relation to episodes of sudden onset of sleep already in 2000 which resulted in special warnings of somnolence and sudden sleep attacks in the non-ergot dopamine agonists' summary of product characteristics.

Beneficial effects of piribedil on parameters of vigilance and cognition have been described in several studies. But, as it seems, no study has been performed so far to identify such effects in the setting of a comparative study with different oral non-ergot dopamine agonists in patients with PD, and utilizing vigilance and cognitive parameters as primary and main secondary objective. The neuropsychological tests being applied in this study are validated and routinely used tests in studies investigating different aspects of attention or vigilance and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian patients aged 35 to 80 years;
* Patients with idiopathic Parkinson's disease;
* Hoehn & Yahr stages 1 to 4;
* Stable medication with anti-parkinsonian medication, including stable treatment with pramipexole or ropinirole, for at least 4 weeks prior to Screening;
* Significant daytime sleepiness: Epworth Sleepiness Scale score equals or is higher than 11 under previous therapy with pramipexole or ropinirole;
* Patients who have read and understood the patient information sheet and have provided a signed written informed consent form;
* Patients are considered to be compliant to the study regimen.

Exclusion Criteria:

* Treatment of Parkinson's disease with any dopamine agonist other than pramipexole or ropinirole within 4 weeks prior to Screening;
* Known hypersensitivity to Clarium® or its excipients;
* Patients with daytime sleepiness caused by other factor's than Parkinson's disease, i.e., idiopathic narcolepsy, shift work, severe alcohol abuse, obstructive diseases, sleep apnea syndrome, or Periodic limb movement disorder;
* Secondary and atypical Parkinson syndrome;
* Depression (Beck Depression Inventory score higher than 16);
* Dementia (Mini-Mental State Examination score equals or is lower than 24);
* Severe disability in extremities which could influence clinical assessments;
* Clinically significant disease concerning the lung, liver or kidney;
* Any acute or chronic infection that may influence the outcome of the study;
* Cardiovascular shock;
* Acute myocardial infarction;
* Congestive heart failure NYHA class III or IV;
* Uncontrolled arterial hypertension (diastolic blood pressure equals or is higher than 105 mmHg) or clinically relevant hypotension;
* Evidence of clinically active cancer;
* Color vision defect that may have impact on assessment of FWIT;
* History of substance abuse;
* Intake of benzodiazepines (or derivates) if not at stable dose for at least 4 weeks prior to Screening; intake of antiallergic agents (H1 receptor antagonists, except selective, non-sedating H1-antihistamines, e.g. loratadine and others), substances with psychostimulant properties (e.g., amphetamine, modafinil), or antidepressants if not at stable dose for at least 2 months prior to Screening;
* Current treatment with neuroleptic agents (except for clozapine);
* Female patients who are pregnant or lactating;
* Female patients of childbearing potential who do not use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly), e.g., implants, injectables, combined oral contraceptives in combination with a barrier method, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner;
* Mental condition rendering the patient unable to understand the nature, scope and possible risks of the study;
* Patient has a history of or is suspicious of unreliability, poor co-operation or non-compliance with medical treatment;
* Patients are currently or previously (within the last 28 days) participating in another study of an investigational drug;
* Patients who were previously enrolled in this study;
* Patients with known Hepatitis B or C or HIV infection;
* Patients who are employees of the sponsor or patients who are employees or relatives of the investigator.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the 'median reaction time during the second 15 minutes (minutes 16-30)' of the subtest 'vigilance', visual test condition 'moving bar', of the Test battery for Attention Performances (TAP) at end of treatment. | Baseline and End of Treatment

SECONDARY OUTCOMES:
Other vigilance parameters of the TAP test | Baseline and End of Treatment
Other neuropsychological tests: Test of verbal fluency (RWT), Verbal learning memory test (VLMT), Stroop test (FWIT) | Baseline and End of Treatment
Epworth Sleepiness Scale (ESS) | Baseline and End of Treatment
Parkinson's Disease Sleeping Scale (PDSS) | Baseline and End of Treatment
Unified Parkinson's Disease Rating Scale (UPDRS) subscores I to IV and total score | Baseline and End of Treatment
Parkinson's disease quality of life questionnaire (PDQ-39) | Baseline and End of Treatment
Clinical Global Impressions (CGI) (except item 3.2) | End of Treatment
Patient Global Impression (PGI) | End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martina Wangemann, Dr., Study Director — Desitin Arzneimittel GmbH
Locations (11):
- Germany (11):
  - Ulm, Baden-Wurttemberg
  - Wolfach, Baden-Wurttemberg
  - München, Bavaria
  - Marburg, Hesse
  - Göttingen, Lower Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
  - Steglitz, State of Berlin
  - Gera, Thuringia
  - Stadtroda, Thuringia